CLINICAL TRIAL: NCT00404157
Title: A Phase III, Extension Study to Evaluate the Safety of Rituximab Retreatment in Subjects With ISN/RPS 2003 Class III or IV Lupus Nephritis Previously Enrolled in Study U2970g
Brief Title: A Study to Evaluate the Safety of Rituximab Retreatment in Subjects With Lupus Nephritis Previously Enrolled in Study U2970g
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: U3388g
Record Dates: First submitted 2006-11-22; First posted 2006-11-27 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Lupus Nephritis
Keywords: Lupus; U2970g
MeSH Terms: conditions — Lupus Nephritis | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab

SUMMARY:
This is a Phase III, multicenter, extension study to evaluate the safety of rituximab administered on a scheduled basis approximately every 6 months. All subjects who complete their Week 52 visit in Study U2970g will be eligible for this study, as long as the inclusion and exclusion criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent and comply with the requirements of the study protocol
* Participation in Study U2970g and completion of the Week 52 visit in that study
* For subjects of reproductive potential (males and females), use of a reliable means of contraception throughout their study participation

Exclusion Criteria:

* Discontinuation or withdrawal from Study U2970g or failure to complete the Week 52 visit
* Any safety concern potentially attributable to rituximab that in the investigator's opinion may jeopardize subject safety
* In the investigator's opinion, lack of any clinical improvement by Week 52 in Study U2970g and for whom the proposed therapy would represent risk without benefit
* Current thrombocytopenia or at high risk for developing clinically significant bleeding or organ dysfunction requiring therapies such as plasmapheresis or acute blood or platelet transfusions
* Lack of peripheral venous access
* Pregnancy or lactation
* History of severe, allergic, or anaphylactic reactions to humanized or murine monoclonal antibodies
* Significant new or uncontrolled disease in any organ system not related to SLE (e.g., poorly controlled chronic obstructive pulmonary disease or asthma, cardiovascular disease, accelerated hypertension, major depression) that in the investigator's opinion would preclude subject participation
* Known active infection of any kind (excluding fungal infection of nail beds), any major episode of infection requiring hospitalization, or treatment with IV antibiotics within 4 weeks of a study drug infusion or oral antibiotics within 2 weeks of a study drug infusion
* History of cancer, including solid tumors, hematologic malignancies, and carcinoma in situ
* Major surgery within 4 weeks prior to screening
* Intolerance or contraindication to oral or IV corticosteroids
* Lipase > 2 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 x the ULN
* Amylase levels > 2 x the ULN
* Absolute neutrophil counts < 1.5 x 10^3/uL
* History of positive hepatitis B surface antigen or hepatitis C serology
* Hemoglobin < 7 g/dL unless caused by autoimmune hemolytic anemia resulting from SLE
* Platelet count < 10,000/uL
* Receipt of a live vaccine within 28 days prior to treatment

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Safety will be monitored through regular physical examinations, vital signs, hematologic laboratory tests, urinalyses, and incidence and severity of adverse events.

SECONDARY OUTCOMES:
Proportion of subjects who maintain a CRR achieved at Week 52 in Study U2970g
Serum rituximab levels
Circulating B-cell counts.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Garg, M.D., Study Director — Genentech, Inc.